CLINICAL TRIAL: NCT04103866
Title: Pressure Offloading Injectible System With the Use of Juvederm Voluma in the Foot
Acronym: POIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Schoenhaus, Jodi, DPM (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POIS Study 1
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-05

CONDITIONS: Metatarsalgia; Hyperkeratotic Callus; Corns; Fat Pad Syndrome
MeSH Terms: conditions — Metatarsalgia; Callosities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pressure Offloading Innersole System (Experimental): Use of Juvederm Voluma in the foot for fat pad restoration
  Interventions: Device: Juvederm Voluma

INTERVENTIONS:
Device: Juvederm Voluma — Juvederm will be used in various parts of the foot to increase collagen volume and decrease high pressures of stress typically seen as people age. It will serve to promote the following: foot cushioning due to tissue atrophy, increase comfort when walking, decrease gait peak pressures which will decrease stress on bones and soft tissue and heal calluses, skin lesions, etc. It will also decrease the patient need for balancing and offloading by the use of an in-shoe orthotic device that requires a closed shoe system. Many people complain of pain walking barefoot, in high heels and sandals where orthotics are not effective.

SUMMARY:
The current use of Juvederm Voluma XC is indicated for deep (subcutaneous and/or supraperiosteal) injection for cheek augmentation to correct age-related volume deficit in the mid-face in adults over the age of 21. In this particular setting, the intended use of the product Juvederm Voluma XC is to show that the filler works to alleviate stress in high pressure areas in the foot during gait, thus decreasing foot pain and allowing individuals to walk more comfortably.

ELIGIBILITY:
Inclusion Criteria:

* Patient's 40 to 75 years of age
* Foot and ankle disability index of at least 55 (based on the majority of people having moderate difficulty in weight-bearing living) and heavy clinical significance of fat atrophy as evaluated by the principal investigator creating a standard analysis.
* Atrophy of the heel or the ball of the foot will be evaluated in the step wise approach.
* Second a clinical exam by the primary investigator

Exclusion Criteria:

* Patients who do not have high pressure fat pad atrophy
* Patient is being treated for cancer
* Skin infections
* Unhealed or acute foot fractures
* Patients with a decrease in dorsalis pedis or posterior tibial pulses
* Pregnant or breast-feeding
* Patients who have had previous injections with fillers
* Patients with nerve injury or nerve damage to the foot causing symptoms of numbness, tingling, burning, and sharp shooting or stabbing sensations. This criteria shall be determined by a. direct patient feedback. If the patient verbally states that they have numbness tingling burning sharp shooting or stabbing pains in their feet or ankles they will not be included.

  b. Semmes Weinstein Monofilament Testing - Semmes Weinstein monofilament testing will be performed on all patients. The Semmes Weinstein will be performed on the great toe submetatarsal one submetatarsal three submetatarsal five the heel and the dorsum of the foot. If a patient cannot feel the sends Weinstein filament in any of those locations they will be eliminated.
* Active an acute diabetic foot ulceration
* Patients with severe allergies manifested by history of anaphylaxis
* Patients with a history or presence of multiple severe allergies
* Patients with a history of allergies to gram-positive bacterial proteins
* Patients with a history of allergies to lidocaine.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
AOFAS | 12 weeks
  The primary endpoint is 12 weeks post injection. The endpoint will be evaluated by the foot and ankle outcome questionnaire for improvement of pain scale scores and ability to return to activity. An improvement that is statistically relevant will be considered an overall total improvement

SECONDARY OUTCOMES:
Less pressure | 52 weeks
  Follow up evaluations: week two, week 24, and week 52. Follow-up evaluation includes: gate pressure mapping with an improvement being a statistically relevant improvement in peek pressure scores before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Foot, Ankle & Leg Vein Center, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided